CLINICAL TRIAL: NCT04816643
Title: A PHASE 1, OPEN-LABEL DOSE-FINDING STUDY TO EVALUATE SAFETY, TOLERABILITY, AND IMMUNOGENICITY AND PHASE 2/3 PLACEBO-CONTROLLED, OBSERVER-BLINDED SAFETY, TOLERABILITY, AND IMMUNOGENICITY STUDY OF A SARS-COV-2 RNA VACCINE CANDIDATE AGAINST COVID-19 IN HEALTHY CHILDREN
Brief Title: A Phase 1/2/3 Study to Evaluate the Safety, Tolerability, and Immunogenicity of an RNA Vaccine Candidate Against COVID-19 in Healthy Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C4591007; 2020-005442-42 (EudraCT Number)
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: SARS-CoV-2 Infection, COVID-19
Keywords: COVID-19; Coronavirus Vaccine; SARS-CoV-2; RNA Vaccine; mRNA Vaccine
MeSH Terms: conditions — COVID-19 | interventions — Biological Products; BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (21):
- Low/Mid-Dose, ≥5 to <12 Years (Experimental): Low/Mid-Dose (10mcg), 2 doses 21 days apart
  Interventions: Biological: Biological/Vaccine: BNT162b2 10mcg
- Mid-Dose, ≥5 to <12 Years (Experimental): Mid-Dose, (20mcg), 2 doses 21 days apart
  Interventions: Biological: BNT162b2 20mcg
- High-Dose, ≥5 to <12 Years (Experimental): High-Dose (30mcg), 2 doses 21 days apart
  Interventions: Biological: BNT162b2 30mcg
- Low/Mid-Dose, ≥2 to < 5 Years (Experimental): Low/Mid-Dose (10mcg), 2 doses 21 days apart
  Interventions: Biological: Biological/Vaccine: BNT162b2 10mcg
- Mid-Dose, ≥2 to <5 Years (Experimental): Mid-Dose, (20mcg), 2 doses 21 days apart
  Interventions: Biological: BNT162b2 20mcg
- High-Dose, ≥2 to <5 Years (Experimental): High-Dose, (30mcg), 2 doses 21 days apart
  Interventions: Biological: BNT162b2 30mcg
- Low/Mid-Dose, ≥6 Months to <2 Years (Experimental): Low/Mid-Dose, (10mcg), 2 doses 21 days apart
  Interventions: Biological: Biological/Vaccine: BNT162b2 10mcg
- Mid-Dose, ≥6 Months to <2 Years (Experimental): Mid-Dose, (20mcg), 2 doses 21 days apart
  Interventions: Biological: BNT162b2 20mcg
- High-Dose, ≥6 Months to <2 Years (Experimental): High-Dose, (30mcg), 2 doses 21 days apart
  Interventions: Biological: BNT162b2 30mcg
- Placebo, ≥6 Months to <2 Years (Placebo Comparator)
  Interventions: Other: Placebo
- Placebo, ≥2 to <5 Years (Placebo Comparator)
  Interventions: Other: Placebo
- Placebo, ≥5 to <12 Years (Placebo Comparator)
  Interventions: Other: Placebo
- Low-Dose, ≥6 Months to <2 Years (Experimental): Low-Dose (3mcg), 2 doses 21 doses apart
  Interventions: Biological: Biological/Vaccine: BNT162b2 3mcg
- Low-Dose, ≥2 to <5 Years (Experimental): Low-Dose (3mcg), 2 doses 21 days apart
  Interventions: Biological: Biological/Vaccine: BNT162b2 3mcg
- High-Dose, 12 to <16 Years (Troponin I Testing) (Experimental): High-Dose (30mcg), 3 doses
  Interventions: Biological: BNT162b2 30mcg
- Low/Mid-Dose, ≥5 to <12 Years (Troponin I Testing) (Experimental): Low/Mid-Dose (10mcg), 3 doses
  Interventions: Biological: Biological/Vaccine: BNT162b2 10mcg
- Placebo, ≥5 to <12 Years (Troponin I Testing) (Experimental)
  Interventions: Other: Placebo
- Low-Dose, ≥6 Months to <2 Years (3-dose regimen) (Experimental): Low-Dose (3mcg), 3 doses
  Interventions: Biological: Biological/Vaccine: BNT162b2 3mcg
- Low-Dose, ≥2 to <5 Years (3-dose regimen) (Experimental): Low-Dose (3mcg), 3 doses
  Interventions: Biological: Biological/Vaccine: BNT162b2 3mcg
- Placebo, ≥6 Months to <2 Years (3-dose regimen) (Placebo Comparator)
  Interventions: Other: Placebo
- Placebo, ≥2 to <5 Years (3-dose regimen) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Biological/Vaccine: BNT162b2 10mcg — BNT162b2 Low/Mid-Dose (10mcg) level
  Arms: Low/Mid-Dose, ≥2 to < 5 Years; Low/Mid-Dose, ≥5 to <12 Years; Low/Mid-Dose, ≥5 to <12 Years (Troponin I Testing); Low/Mid-Dose, ≥6 Months to <2 Years
Biological: BNT162b2 20mcg — BNT162b2 Mid-Dose (20mcg) level
  Arms: Mid-Dose, ≥2 to <5 Years; Mid-Dose, ≥5 to <12 Years; Mid-Dose, ≥6 Months to <2 Years
Biological: BNT162b2 30mcg — BNT162b2 High-Dose (30mcg) level
  Arms: High-Dose, 12 to <16 Years (Troponin I Testing); High-Dose, ≥2 to <5 Years; High-Dose, ≥5 to <12 Years; High-Dose, ≥6 Months to <2 Years
Other: Placebo — Intramuscular injection
  Arms: Placebo, ≥2 to <5 Years; Placebo, ≥2 to <5 Years (3-dose regimen); Placebo, ≥5 to <12 Years; Placebo, ≥5 to <12 Years (Troponin I Testing); Placebo, ≥6 Months to <2 Years; Placebo, ≥6 Months to <2 Years (3-dose regimen)
Biological: Biological/Vaccine: BNT162b2 3mcg — BNT162b2 Low-Dose (3mcg) level
  Arms: Low-Dose, ≥2 to <5 Years; Low-Dose, ≥2 to <5 Years (3-dose regimen); Low-Dose, ≥6 Months to <2 Years; Low-Dose, ≥6 Months to <2 Years (3-dose regimen)

SUMMARY:
This is a Phase 1/2/3 study in healthy children.

Dependent upon safety and/or immunogenicity data generated during the course of this study, and the resulting assessment of benefit-risk, the safety, tolerability, and immunogenicity of BNT162b2 in participants <6 months of age may subsequently be evaluated.

DETAILED DESCRIPTION:
Phase 1 Dose-Finding

Is the open-label dose-finding portion of the study that will evaluate safety, tolerability, and immunogenicity of BNT162b2 administered on a 2-dose (separated by approximately 21 days) schedule in up to 3 age groups (participants ≥5 to <12 years, ≥2 to <5 years, and ≥6 months to <2 years of age).

Dose finding is being initiated in this study in participants ≥5 to <12 years of age based on the acceptable blinded safety assessment of the 30-µg dose in 12- to 15-year-olds in the C4591001 study.

The purpose of Phase 1 is to identify preferred dose level(s) of BNT162b2 from up to 3 different dose levels in each age group.

Dependent upon safety and/or immunogenicity data generated during the course of this study, it is possible that dose levels may not be started, may be terminated early, and/or may be added with dose levels below the lowest stated dose.

Update as part of protocol amendment 6: All participants will receive a third dose of BNT162b2. For participants ≥6 months to <5 years, the third dose will occur at least 8 weeks after the second dose. In participants ≥5 to <12 years, the third dose will occur at least 6 months after the second dose. The interval between the second and third doses will be based on the participant's age at the time of enrollment. The dose level of the third dose of BNT162b2 will be based on age at the time of vaccination: participants <5 years of age at the time of the third dose will receive the 3-µg dose level, participants ≥5 to <12 years of age at the time of the third dose will receive the 10-µg dose level, and participants ≥12 years of age at the time of the third dose will receive the 30-µg dose level.

Participants will have blood drawn prior to both Dose 1 and Dose 2 and 7 days after Dose 2 to assess immunogenicity to determine the selected BNT162b2 dose level for Phase 2/3. Participants will also have blood drawn prior to Dose 3 and 1, 6, and 12 months after Dose 3.

Phase 2/3 Selected-Dose

Is the portion of the study that will evaluate the safety, tolerability, and immunogenicity in each age group at the selected dose level from the Phase 1 dose-finding portion of the study. Efficacy will be evaluated within or across age groups in which immunobridging is successful, depending on accrual of a sufficient number of cases in those age groups.

Participants will have blood drawn at baseline prior to Dose 1 and 6 months after Dose 2. Immunobridging to participants 16 to 25 years of age in the C4591001 study will be based on immunogenicity data collected at (1) baseline and 1 month after Dose 2 and (2) baseline and 1 month after Dose 3. The persistence of the immune response will be based on immunogenicity data collected in participants at (1) baseline and 1 and 6 months after Dose 2 and (2) baseline and 1, 6, 12, and 18 months after Dose 3. In addition, efficacy against confirmed COVID-19 and against asymptomatic infection will also be assessed in participants ≥5 to <12 years of age.

At designated US sites, an additional optional whole blood sample of approximately 10 mL will be obtained prior to Dose 1 and at 7 days and 6 months after Dose 2 from up to approximately 60 participants ≥10 years of age. Additional samples will be obtained prior to Dose 3 and 1 month after Dose 3 (original BNT162b2 group only). These samples will be used on an exploratory basis to investigate the postvaccination cell-mediated immune response at these time points.

At the 6-month follow-up visit, all participants will be unblinded. Participants who originally received placebo will be offered the opportunity to receive BNT162b2 as part of the study. Participants who originally received placebo and become eligible for receipt of BNT162b2 or another COVID-19 vaccine according to local or national recommendations prior to the 6 month follow-up visit (Visit 5 or 405) (detailed separately and available in the electronic study reference portal) will have the opportunity to receive BNT162b2 (10 µg or 3 µg) based on age at the time of vaccination.

Update as part of protocol amendment 6: All participants will receive a third dose of BNT162b2. For participants ≥6 months to <5 years, the third dose will occur at least 8 weeks after the second dose. In participants ≥5 to <12 years, the third dose will occur at least 6 months after the second dose. The interval between the second and third doses will be based on the participant's age at the time of enrollment. The dose level of the second and third doses of BNT162b2 will be based on age at the time of vaccination: participants <5 years of age at the time of the second/third dose will receive the 3-µg dose level, participants ≥5 to <12 years of age at the time of the second/third dose will receive the 10-µg dose level, and participants ≥12 years of age at the time of the second/third dose will receive the 30-µg dose level.

Phase 2/3 Obtaining Serum Samples for Potential Troponin I Testing

If testing of troponin I levels in individuals who did not receive BNT162b2 indicates that troponin I level could be a reliable indicator of potential subclinical myocarditis, obtaining serum samples for potential troponin I testing during the period of increased risk of clinical myocarditis may help characterize the absence/presence and frequency of subclinical myocarditis. To assess, an additional group of participants will be included: ≥5 to <12 years: randomized 2:1 to receive BNT162b2 10 µg or placebo, and ≥12 to <16 years of age: open-label receipt of BNT162b2 30 µg.

Update as part of protocol amendment 7: All participants will receive a third dose of BNT162b2. For all participants (≥5 to <12 and ≥12 to <16 years of age), the third dose will occur at least 5 months after Dose 2.

The dose level of the second and third doses of BNT162b2 will be based on age at the time of vaccination: participants ≥5 to <12 years of age at the time of the second/third dose will receive the 10-µg dose level, and participants ≥12 years of age at the time of the second/third dose will receive the 30-µg dose level.

Update as part of protocol amendment 8: The Lower-Dose Evaluation portion of the protocol has been removed.

Participation in the study will cease 6 months after the third dose of BNT162b2.

ELIGIBILITY:
Inclusion Criteria

1. Male or female participants ≥6 months to <12 years of age, at the time of randomization, at Visit 1 for the dose-finding/selected-dose evaluation. For the obtaining-serum-samples-for-potential-troponin I-testing portion of the study: Male or female participants between ≥5 and <16 years of age.
2. Participants' parent(s)/legal guardian(s) and participants, as age appropriate, who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
3. Healthy participants who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.

   Note: Healthy participants with preexisting stable disease, defined as disease not requiring significant change in the therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included.
4. Participants are expected to be available for the duration of the study and whose parent(s)/legal guardian can be contacted by telephone during study participation.
5. Negative urine pregnancy test for female participants who are biologically capable of having children.
6. Female participant of childbearing potential or male participant able to father children who is willing to use a highly effective method of contraception as outlined in this protocol for at least 28 days after the last dose of study intervention if at risk of pregnancy with her/his partner; or female participant not of childbearing potential or male participant not able to father children.
7. The participant or participant's parent(s)/legal guardian is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol. Depending on the age of the participant and according to local requirements, participants will also be asked to provide assent as appropriate (verbal or written).

Exclusion Criteria

1. Phase 1 only: Past clinical (based on COVID-19 symptoms/signs alone, if a SARS CoV 2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID 19.
2. Phase 1 only: Known infection with HIV, HCV, or HBV.
3. Receipt of medications intended to prevent COVID-19.
4. Previous or current diagnosis of MIS-C.
5. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study. Note: This includes both conditions that may increase the risk associated with study intervention administration or a condition that may interfere with the interpretation of study results
6. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
7. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
8. Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic lupus erythematosus. Note: Stable type 1 diabetes and hypothyroidism are permitted.
9. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
10. Female who is pregnant or breastfeeding.
11. Previous vaccination with any coronavirus vaccine.
12. Individuals who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
13. Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19 from 90 days before study intervention administration, or planned receipt throughout the study.
14. Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
15. Previous participation in other studies involving study intervention containing LNPs.
16. Participants who are direct descendants (child or grandchild) of investigational site staff members or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11837 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Percentage of participants in Phase 1 reporting local reactions | for 7 days after Dose 1 and Dose 2
  Pain or tenderness at the injection site, redness and swelling as reported on electronic diaries.
Percentage of participants in Phase 1 reporting systemic events | for 7 days after Dose 1 and Dose 2
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened join pain, decreased appetite drowsiness, and irritability as reported on electronic diaries
Percentage of participants in Phase 1 reporting adverse events | from Dose 1 through 1 month after the last dose
  As elicited by investigational site staff
Percentage of participants in Phase 1 reporting serious adverse events | from Dose 1 through 6 months after the last dose
  As elicited by investigational site staff
Percentage of participants in Phase 2/3 reporting local reaction | for 7 days after Dose 1 and Dose 2
  Pain or tenderness at the injection site, redness and swelling as reported on electronic diaries.
Percentage of participants in Phase 2/3 reporting systemic events | for 7 days after Dose 1 and Dose 2
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, new or worsened joint pain, decreased appetite, drowsiness, and irritability as reported on electronic diaries
Percentage of participants in Phase 2/3 reporting adverse events | from Dose 1 through 1 month after the last dose
  As elicited by investigational site staff
Percentage of participants in Phase 2/3 reporting serious adverse events | from Dose 1 through 6 months after the last dose
  As elicited by investigational site staff
Ph 2/3 selected-dose (2-dose series), immunobridging of SARS-CoV-2 serum neutralizing titers after 2 doses in participants ≥5 to <12 years to the geometric mean of SARS-CoV-2 serum neutralizing titers in participants 16 to 25 years in the C4591001 study | 1 month after the second dose
  As measured at the central laboratory
Ph 2/3 selected-dose (2-dose series), immunobridging of SARS-CoV-2 serum neutralizing titers after 2 doses in participants ≥2 to <5 years to the geometric mean of SARS-CoV-2 serum neutralizing titers in participants 16 to 25 years in the C4591001 study | 1 month after the second dose
  As measured at the central laboratory
Ph 2/3 selected-dose (2-dose series), immunobridging of SARS-CoV-2 serum neutralizing titers after 2 doses in participants ≥6 months to <2 years to the geometric mean of SARS-CoV-2 serum neutralizing titers in participants 16 to 25 in C4591001 study | 1 month after the second dose
  As measured at the central laboratory
In Phase 2/3 selected-dose (2-dose series), the difference in percentages of participants with seroresponse in participants ≥5 to <12 years of age and participants 16 to 25 years of age from Phase 2/3 of the C4591001 study | 1 month after the second dose
  As measured at the central laboratory
In Phase 2/3 selected-dose (2-dose series), the difference in percentages of participants with seroresponse in participants ≥2 to <5 years of age and participants 16 to 25 years of age from Phase 2/3 of the C4591001 study | 1 month after the second dose
  As measured at the central laboratory
In Phase 2/3 selected-dose (2-dose series), the difference in percentages of participants with seroresponse in participants ≥6 months to <2 years of age and participants 16 to 25 years of age from Phase 2/3 of the C4591001 | 1 month after the second dose
  As measured at the central laboratory
Ph 2/3 selected-dose (3-dose series), immunobridging of SARS-CoV-2 serum neutralizing titers after 3 doses in participants ≥2 to <5 years to the geometric mean of SARS-CoV-2 serum neutralizing titers in C4591001 participants 16 to 25 years after 2 doses | 1 month after the third dose
  As measured at the central laboratory
Ph 2/3 selected-dose (3-dose), immunobridging SARS-CoV-2 serum neutralizing titers after 3 doses in participants ≥6 months to <2 years to the geometric mean of SARS-CoV-2 serum neutralizing titers in C4591001 participants 16 to 25 in study after 2 doses | 1 month after the third dose
  As measured at the central laboratory
In Phase 2/3 selected-dose (3-dose series), the difference in percentages of participants with seroresponse in participants ≥2 to <5 years of age and participants 16 to 25 years of age from Phase 2/3 of the C4591001 study | 1 month after the third dose
  As measured at the central laboratory
In Phase 2/3 selected-dose (3-dose series), the difference in percentages of participants with seroresponse in participants ≥6 months to <2 years of age and participants 16 to 25 years of age from Phase 2/3 of the C4591001 | 1 month after the third dose
  As measured at the central laboratory

SECONDARY OUTCOMES:
In Phase 1 participants, SARS-CoV-2 serum neutralizing antibody levels, expressed as GMTs | At each time point
  As measured at the central laboratory
In evaluable Phase 2/3 participants at selected dose level in each age group, Geometric Mean Titers of SARS-CoV-2 neutralizing titers with no serological or virological evidence of past SARS-CoV-2 infection | At baseline (before Dose 1) and 1, 6, 12 (for the original BNT162b2 group only), and 24 (for the original BNT162b2 group only) months after Dose 2
  As measured at the central laboratory
In evaluable Phase 2/3 participants at the dose level selected in each age group, Geometric Mean Fold Ratio in SARS-CoV-2 serum neutralizing titer from before vaccination to each subsequent time point | From before Dose 1 to each subsequent time point after Dose 2
  As measured at the central laboratory
Ratio of confirmed COVID-19 illness, Phase 2/3 selected-dose participants ≥5 to <12 years of age with successful immunobridging, without evidence of prior SARS-CoV-2 infection for the active vaccine group to the placebo group | From 7 days after the second dose to prior to third dose
  Per 1000 person-years of follow-up
Ratio of confirmed COVID-19 illness, Phase 2/3 selected-dose participants ≥5 to <12 years of age with successful immunobridging, with and without evidence of prior SARS-CoV-2 infection for the active vaccine group to the placebo group | From 7 days after the second dose to prior to third dose
  Per 1000 person-years of follow-up
Ratio of confirmed COVID-19 illness, Phase 2/3 selected-dose participants ≥6 months to <5 years of age (3-dose series), evidence of prior SARS-CoV-2 infection for the active vaccine group to the placebo group | From 7 days after the third dose
  1000 person-years of follow-up
Ratio of confirmed COVID-19 illness, Phase 2/3 selected-dose participants ≥6 months to <5 years of age (3-dose series), with and without evidence of prior SARS-CoV-2 infection for the active vaccine group to the placebo group | From 7 days after the third dose
  1000 person-years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (144):
- United States (98):
  - University of Alabama at Birmingham - School of Medicine, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - SCPMG/Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Matrix Clinical Research, Los Angeles, California
  - Madera Family Medical Group, Madera, California
  - Kaiser Permanente Oakland, Oakland, California
  - Clinical & Translational Research Unit (CTRU) & Spectrum BioBank, Stanford University, Palo Alto, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Center for Clinical Trials, Paramount, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Kaiser Permanente Sacramento, Sacramento, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Stanford Health Care Investigational Drug Service, Stanford, California
  - Stanford Health Care, Stanford, California
  - Bayview Research Group, LLC, Valley Village, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Emerson Clinical Research Institute - Washington - Connecticut Avenue, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Meridian Clinical Research, LLC, Washington D.C., District of Columbia
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Emory Children's Center Illness POD, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Meridian Clinical Research, LLC, Macon, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Novak Center for Children's Health, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana State University Health Sciences Shreveport, Shreveport, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Michigan Center of Medical Research, Bingham Farms, Michigan
  - Quinn Healthcare/SKYCRNG, Ridgeland, Mississippi
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Meridian Clinical Research, LLC, Hastings, Nebraska
  - Velocity Clinical Research, Lincoln, Lincoln, Nebraska
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - Children's Physician's Clinic, Spring Valley, Omaha, Nebraska
  - Rutgers University, New Brunswick, New Jersey
  - Meridian Clinical Research LLC, Binghamton, New York
  - Meridian Clinical Research, LLC, Binghamton, New York
  - Advanced Specialty Care, Commack, New York
  - Clinical Research Center, East Setauket, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Atrium Health-STRIVE Vaccine Research Clinic, Charlotte, North Carolina
  - Teen Health Connection (study visits), Charlotte, North Carolina
  - Duke University - Main Hospital and Clinics, Durham, North Carolina
  - Duke Vaccine And Trials Unit, Durham, North Carolina
  - Atrium Health-STRIVE Vaccine Research Clinic (study visits), Matthews, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - AHN Erie Health + Wellness Pavillion: West, Erie, Pennsylvania
  - Velocity Clinical Research-Providence, East Greenwich, Rhode Island
  - Coastal Pediatric Research, Charleston, South Carolina
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Coastal Pediatric Research, Summerville, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Clinical Research Associates Inc, Nashville, Tennessee
  - ARC Clinical Research at Four Points, Austin, Texas
  - ARC Clinical Research at Wilson Parke, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Cedar Health Research, Dallas, Texas
  - Bay Colony Pediatrics, Dickinson, Texas
  - Proactive Clinical Research, LLC, Edinburg, Texas
  - Village Health Partners (Patient Seen Address), Frisco, Texas
  - Helios Clinical Research - HOU, Houston, Texas
  - Van Tran Family Practice, Houston, Texas
  - Texas Children's Hospital - Clinical Research Center, Houston, Texas
  - West Houston Clinical Research Services, Houston, Texas
  - DM Clinical Research, Houston, Texas
  - Pediatric Associates, Houston, Texas
  - ACRC Trials (Administrative Site), Plano, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Pediatric Associates of Charlottesville, PLC (Private Pediatric Practice), Charlottesville, Virginia
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - Virginia Research Center, Midlothian, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Brazil (5):
  - Hospital Santo Antônio - Obras Sociais Irmã Dulce/ Centro de Pesquisa Clínica - CPEC, Salvador, Estado de Bahia
  - Santa Casa De Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Serviço de Infectologia e Controle de Infecção Hospitalar de Curitiba/ Centro Médico São Franci, Curitiba, Paraná
  - CePCLIN - Centro de Estudos e Pesquisas em Moléstias Infecciosas Ltda, Natal, Rio Grande do Norte
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos Ltda., São Paulo
- Finland (14):
  - FVR, Oulu Clinic, Oulu, North Ostrobothnia
  - Tampere Vaccine Research Clinic, Tampere, Pirkanmaa
  - FVR, Helsinki East Clinic, Helsinki, Southwest Finland
  - FVR, Helsinki East Clinic, Helsinki, Uusimaa
  - FVR, Järvenpää Clinic, Jarvenpaa, Uusimaa
  - FVR, Espoo Clinic, Espoo
  - FVR, Helsinki South Clinic, Helsinki
  - MeVac - Meilahti Vaccine Research Center, Helsinki
  - FVR, Helsinki East Clinic, Helsinki
  - FVR, Kokkola Clinic, Kokkola
  - FVR, Pori Clinic, Pori
  - FVR, Seinäjoki Clinic, Seinäjoki
  - FVR, Tampere Clinic, Tampere
  - FVR, Turku Clinic, Turku
- Mexico (4):
  - CHRISTUS - LATAM HUB Center of excellence and innovation S.C., Monterrey, Nuevo León
  - Kohler & Milstein Research S.A. de C.V., Mérida, Yucatán
  - Centro Multidisciplinario Para El Desarrollo Especializado De La Investigacion, Mérida, Yucatán
  - Sociedad de Metabolismo y Corazón S.C., Veracruz
- Poland (8):
  - MICS Centrum Medyczne Torun, Torun, Kuyavian-Pomeranian Voivodeship
  - IN-VIVO Bydgoszcz, Bydgoszcz
  - Centrum Badan Klinicznych JCI, Krakow
  - Osrodek Badan Klinicznych Appletreeclinics, Lodz
  - GRAVITA Diagnostyka i Leczenie nieplodnosci, Lodz
  - Rodzinne Centrum Medyczne LUBMED, Luboń
  - Niepubliczny Zaklad Lecznictwa Ambulatoryjnego Michalkowice Jarosz i Partnerzy Spolka Lekarska, Siemianowice Śląskie
  - Provita 001, Warsaw
- Spain (15):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruna
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, A Coruña
  - EAP Centelles, Centelles, Barcelona
  - EBA Centelles, Centelles, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregrat, Barcelona
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Hospital Universitario HM Puerta del Sur, Madrid, Madrid, Comunidad de
  - Hospital de Antequera, Antequera, Malaga
  - Hospital de Antequera, Antequera, Málaga
  - Grupo Pediatrico Uncibay, Málaga, Málaga
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital HM Puerta del Sur, Móstoles
  - Instituto Hispalense de Pediatria, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pather S, Charpentier N, van den Ouweland F, Rizzi R, Finlayson A, Salisch N, Muik A, Lindemann C, Khanim R, Abduljawad S, Smith ER, Gurwith M, Chen RT; Benefit-Risk Assessment of VAccines by TechnolOgy Working Group (BRAVATO; ex-V3SWG). A Brighton Collaboration standardized template with key considerations for a benefit-risk assessment for the Comirnaty COVID-19 mRNA vaccine. Vaccine. 2024 Sep 17;42(22):126165. doi: 10.1016/j.vaccine.2024.126165. Epub 2024 Aug 27. PMID 39197299
- [Derived] Simoes EAF, Klein NP, Sabharwal C, Gurtman A, Kitchin N, Ukkonen B, Korbal P, Zou J, Xie X, Sarwar UN, Xu X, Lockhart S, Cunliffe L, Lu C, Ma H, Swanson KA, Koury K, Shi PY, Cooper D, Tureci Ӧ, Jansen KU, Sahin U, Gruber WC. Immunogenicity and Safety of a Third COVID-19 BNT162b2 mRNA Vaccine Dose in 5- to 11-Year Olds. J Pediatric Infect Dis Soc. 2023 Apr 28;12(4):234-238. doi: 10.1093/jpids/piad015. PMID 36929216
- [Derived] Munoz FM, Sher LD, Sabharwal C, Gurtman A, Xu X, Kitchin N, Lockhart S, Riesenberg R, Sexter JM, Czajka H, Paulsen GC, Maldonado Y, Walter EB, Talaat KR, Englund JA, Sarwar UN, Hansen C, Iwamoto M, Webber C, Cunliffe L, Ukkonen B, Martinez SN, Pahud BA, Munjal I, Domachowske JB, Swanson KA, Ma H, Koury K, Mather S, Lu C, Zou J, Xie X, Shi PY, Cooper D, Tureci O, Sahin U, Jansen KU, Gruber WC; C4591007 Clinical Trial Group. Evaluation of BNT162b2 Covid-19 Vaccine in Children Younger than 5 Years of Age. N Engl J Med. 2023 Feb 16;388(7):621-634. doi: 10.1056/NEJMoa2211031. PMID 36791162
- [Derived] Walter EB, Talaat KR, Sabharwal C, Gurtman A, Lockhart S, Paulsen GC, Barnett ED, Munoz FM, Maldonado Y, Pahud BA, Domachowske JB, Simoes EAF, Sarwar UN, Kitchin N, Cunliffe L, Rojo P, Kuchar E, Ramet M, Munjal I, Perez JL, Frenck RW Jr, Lagkadinou E, Swanson KA, Ma H, Xu X, Koury K, Mather S, Belanger TJ, Cooper D, Tureci O, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591007 Clinical Trial Group. Evaluation of the BNT162b2 Covid-19 Vaccine in Children 5 to 11 Years of Age. N Engl J Med. 2022 Jan 6;386(1):35-46. doi: 10.1056/NEJMoa2116298. Epub 2021 Nov 9. PMID 34752019
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591007